CLINICAL TRIAL: NCT02846116
Title: Evaluation of Patient Satisfaction and Shade Matching of Vita Suprinity Versus Lithium Disilicate (E-max) Ceramic Crowns in Esthetic Zone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Abou-steit, Principal investigator, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-2016-7-170
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Personal Satisfaction
Keywords: all ceramic crown; Lithium disilicate; e-max; vita suprinity
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lithium disilicate (Active Comparator): The intervention will be: Prosthetic crown
  Interventions: Other: Prosthetic crown
- Vita suprinity (Active Comparator): The intervention will be: Prosthetic crown
  Interventions: Other: Prosthetic crown

INTERVENTIONS:
Other: Prosthetic crown
  Other Names: all ceramic crown

SUMMARY:
The aim of this study is to evaluate using of new ceramic material Vita Suprinity and lithium disilicate on patient satisfaction combined with shade matching.

DETAILED DESCRIPTION:
Justification for undertaking the trial:

Nowadays, esthetics has become an important aspect of dentistry due to decrease in caries prevalence and increase in patients' perception of their teeth appearance. Therefore dentists should take into consideration the esthetic needs of the patients during treatment, otherwise patient satisfaction will not be achieved with its subsequent influence on patient self quality of life and psychological status.

As a survey concerning patient satisfaction with regard to dental esthetics issues concluded that color of the restoration plays a primary role for patient satisfaction, as 89.3% of patients were dissatisfied of their dental appearance because of their restorations' color.

Therefore the use of ceramic crowns has increased substantially in recent years because of their superior esthetics and color rendering. In addition to their ability to achieve complete patient satisfaction.

Rationale:

Achieving good esthetic results especially with the continuous innovations of dental ceramic materials is not always easy to achieve and the definitive shade match of porcelain restorations to natural dentition remains a challenge to the dental practitioners and ceramists. Furthermore patient satisfaction to the final outcome is not always in agreement with the clinicians in regard to shade matching decisions.

Therefore this study will be conducted to evaluate patient satisfaction and shade matching of Vita suprinity versus e-max all ceramic crowns in esthetic zone.

Benefits of the research to the patient:

Patient will receive a restoration with superior esthetics, shade match and quality.

It will provide the patient with long-term predictable esthetic restorations As a result of unnoticed perfect esthetic restoration, the patient will be psychologically improved.

Benefits of the research to the clinician:

Practitioner will have the advantage to assess a new material that can be used in different situations for better esthetic outcomes.

It will improve patient confidence with the dentist. It will improve professional skills of the dentist to achieve optimum esthetic results.

Explanation for choice of comparators:

The use of IPS e.max Press is well documented in the literatures as successful restoration modality. A three-year clinical evaluation of two ceramic crown systems revealed excellent color match for the IPS e-max crowns (Alpha for 24 crowns and Bravo for 6 crowns with slight shade mismatches). Also patient questionnaire revealed satisfaction with the appearance and comfort of their restorations.

A 2 years prospective clinical observation study reported Alpha scores (greater than 92%) indicating no appreciable change in the crowns during the two years of the study.

Also the clinical performance of lithium disilicate pressable ceramic crowns revealed a survival rate of 97.4 % after 5 years and 94.8 % after 8 years as reported by Gehrt et al., (2013).

Another 2 years clinical evaluation of lithium disilicate based all ceramic crowns revealed satisfactory clinical performance, with color match Alpha (85%) at baseline, 80% at 1 year recall and 60 % at 2 years recall.

Research hypothesis:

There is difference in the clinical performance of Vita Suprinity if compared with Lithium disilicate ceramic crown restoration if used in esthetic zone.

Interventions:

VITA SUPRINITY: Vita suprinity product Brochure presented a new generation of glass ceramic material. With the aid of an innovative manufacturing process, the glass ceramic is enriched with approximately 10% zirconia by weight, resulting in the world's first zirconia reinforced lithium silicate ceramic (ZLS). The material features a special fine-grained, homogeneous structure that provides excellent material quality and consistency, high load capacity and long term reliability. Moreover, the material offers natural esthetics with successful outcome. Also it offers outstanding processing characteristics, including easy milling and polishing.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 20-60 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
2. Patients able physically and psychologically to tolerate conventional restorative procedures.
3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
4. Patients with teeth problems indicated for full coverage restoration (e.g. mild to moderate discoloration, coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
5. Patients with root canal treated teeth requiring full coverage restorations.
6. Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with poor oral hygiene and motivation.
3. Pregnant women's to avoid any complication that may occur in dental office due to pregnancy or due to injected anesthetic solution.
4. Patients with psychiatric problems or unrealistic expectation (patient that has phobia from dental treatments or needle bunch).
5. Patients have no opposite occluding dentition in the area intended for restoration.
6. Patients suffer from parafunctional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction using Visual Analogue scale- Binary (Satisfied or not satisfied) | 1 year

SECONDARY OUTCOMES:
Shade matchUsing the modified United States Public Health Service criteria (Modified USPHS)- categorical | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amina Zaki, Professor, Study Director — Faculty of Oral and Dental Medicine- Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tin-Oo MM, Saddki N, Hassan N. Factors influencing patient satisfaction with dental appearance and treatments they desire to improve aesthetics. BMC Oral Health. 2011 Feb 23;11:6. doi: 10.1186/1472-6831-11-6. PMID 21342536
- [Background] Batson ER, Cooper LF, Duqum I, Mendonca G. Clinical outcomes of three different crown systems with CAD/CAM technology. J Prosthet Dent. 2014 Oct;112(4):770-7. doi: 10.1016/j.prosdent.2014.05.002. Epub 2014 Jun 28. PMID 24980739
- [Background] John MT, Slade GD, Szentpetery A, Setz JM. Oral health-related quality of life in patients treated with fixed, removable, and complete dentures 1 month and 6 to 12 months after treatment. Int J Prosthodont. 2004 Sep-Oct;17(5):503-11. PMID 15543905
- [Background] Grossmann AC, Hassel AJ, Schilling O, Lehmann F, Koob A, Rammelsberg P. Treatment with double crown-retained removable partial dentures and oral health-related quality of life in middle- and high-aged patients. Int J Prosthodont. 2007 Nov-Dec;20(6):576-8. PMID 18069364
- [Background] Corciolani G, Vichi A, Louca C, Ferrari M. Color match of two different ceramic systems to selected shades of one shade guide. J Prosthet Dent. 2011 Mar;105(3):171-6. doi: 10.1016/S0022-3913(11)60025-5. PMID 21356409
- [Background] Ishikawa-Nagai S, Yoshida A, Sakai M, Kristiansen J, Da Silva JD. Clinical evaluation of perceptibility of color differences between natural teeth and all-ceramic crowns. J Dent. 2009;37 Suppl 1:e57-63. doi: 10.1016/j.jdent.2009.04.004. Epub 2009 Apr 18. PMID 19423209
- [Background] Al-Wahadni A, Ajlouni R, Al-Omari Q, Cobb D, Dawson D. Shade-match perception of porcelain-fused-to-metal restorations: a comparison between dentist and patient. J Am Dent Assoc. 2002 Sep;133(9):1220-5; quiz 1260-1. doi: 10.14219/jada.archive.2002.0363. PMID 12356253
- [Background] Etman MK, Woolford MJ. Three-year clinical evaluation of two ceramic crown systems: a preliminary study. J Prosthet Dent. 2010 Feb;103(2):80-90. doi: 10.1016/S0022-3913(10)60010-8. PMID 20141812
- [Background] Dr Rupal J Shah1. A Study of Patient Satisfaction with Maxillary Anterior Teeth Restorations and Desirable Esthetic Treatment Options\n. IOSR J. Dent. Med. Sci. 13, 79-86 (2014).
- [Result] Samorodnitzky-Naveh GR, Geiger SB, Levin L. Patients' satisfaction with dental esthetics. J Am Dent Assoc. 2007 Jun;138(6):805-8. doi: 10.14219/jada.archive.2007.0269. PMID 17545270